CLINICAL TRIAL: NCT02361372
Title: Short-term Effect of Kefir-fermented Milk Consumption on Bone Mineral Density and Bone Metabolism in Osteoporotic Patients
Brief Title: Kefir on Bone Mineral Density and Bone Metabolism in Osteoporotic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Min-Yu Tu, Ministry of Science and Technology, Ministry of Science and Technology, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NSC-99-2324-B-005-017-CC1
Record Dates: First submitted 2014-09-26; First posted 2015-02-11 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Kefir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Kefir and CaCO3 (Experimental): Kefir were administered 1,600 mg kefir-fermented milk per day and an accompanying supplement of 1,500 mg CaCO3 for 6 months
  Interventions: Other: Kefir
- Placebo and CaCO3 (Placebo Comparator): Placebo and 1,500 mg of CaCO3 daily for 6 months
  Interventions: Other: Placebo; Other: CaCO3

INTERVENTIONS:
Other: Placebo — Placebo daily for 6 months
  Arms: Placebo and CaCO3
Other: CaCO3 — CaCO3 daily for 6 months
  Arms: Placebo and CaCO3
Other: Kefir — Kefir daily for 6 months
  Arms: Kefir and CaCO3

SUMMARY:
In a controlled, parallel, double-blind intervention study over 6 months, the investigators investigated the effects of kefir-fermented milk (1,600 mg/kg) supplemented with calcium bicarbonate (CaCO3, 1,500 mg/kg) and bone metabolism in 40 osteoporosis patients, and compared them with CaCO3 alone without kefir supplements. Bone turnover markers were measured in fasting blood samples collected before therapy and at 1, 3, and 6 months. BMD values at the spine, total hip, and hip femoral neck were assessed by dual-energy x-ray absorptiometry (DXA) at baseline and at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of osteoporosis patients

Exclusion Criteria:

* Any previous use of parathyroid hormone or sodium fluoride, use of anabolic steroids or growth hormone within 6 months before trial entry or oral or intravenous systemic corticosteroids within 12 months, and any previous use of strontium.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2010-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
bone mineral density and bone regeneration | 3 months

REFERENCES:
- [Derived] Tu MY, Chen HL, Tung YT, Kao CC, Hu FC, Chen CM. Short-Term Effects of Kefir-Fermented Milk Consumption on Bone Mineral Density and Bone Metabolism in a Randomized Clinical Trial of Osteoporotic Patients. PLoS One. 2015 Dec 10;10(12):e0144231. doi: 10.1371/journal.pone.0144231. eCollection 2015. PMID 26655888